CLINICAL TRIAL: NCT03493984
Title: A Preliminary Clinical Trial Investigating the Ability of Plant Exosomes to Mitigate Insulin Resistance and Chronic Inflammation in Patients Diagnosed With Polycystic Ovary Syndrome (PCOS)
Brief Title: Plant Exosomes and Patients Diagnosed With Polycystic Ovary Syndrome (PCOS) 17
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the university prior to study approval, no patients enrolled
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17.1114
Record Dates: First submitted 2018-02-20; First posted 2018-04-11 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ginger exosomes (Experimental)
  Interventions: Other: Ginger exosomes
- Aloe exosomes (Experimental)
  Interventions: Other: Aloe exosomes
- Ginger and aloe exosomes (Experimental)
  Interventions: Other: Ginger exosomes; Other: Aloe exosomes
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ginger exosomes — Naturally occurring plant exosomes from ginger
  Arms: Ginger and aloe exosomes; Ginger exosomes
Other: Aloe exosomes — Naturally occurring plant exosomes from aloe
  Arms: Aloe exosomes; Ginger and aloe exosomes
Other: Placebo — Exosome placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if substances contained in ginger or aloe plants, called exosomes, will treat and improve the condition polycystic ovary syndrome

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 year
* Patients must have a confirmed diagnosis of PCOS according to the Rotterdam Criteria. At least 2 of the following 3 characteristics must be present: 1. Oligo-anovulation 2. Clinical and/or biochemical signs of androgen excess and 3. Polycystic ovarian morphology (PCOM) (defined by an increased number of small antral follicles [≥12 follicles that were <10 mm in diameter] or an increased individual ovarian volume [>10 cm3] in 1 or both ovaries. Disorders mimicking PCOS must also be excluded, including thyroid dysfunction, hyperprolactinemia, late-onset congenital adrenal hyperplasia, and ovarian or adrenal androgen-producing tumors.
* Of all subjects screened patients must be informed of the investigational nature of this study and give written informed consent in accordance with institutional and federal guidelines.
* Ability to understand and willingness to sign a written informed consent document.
* Absence of life limiting medical conditions

Exclusion Criteria:

* • Pregnancy

  * Known HIV
  * Patients receiving immunosuppressive drugs
  * Patients taking confounding medications such as sex steroids, infertility medications or insulin sensitizers or any medication deemed to alter glucose and/or insulin levels
  * Active malignancy in the last 5 years
  * Patients receiving any other investigational agent(s)
  * Ginger and/or aloe allergy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in glucose tolerance as measured by a glucose tolerance test | Baseline, twelve weeks.
  A glucose challenge test will be administered after initially obtaining a fasting serum glucose(baseline), then administering a 75 gram glucose load orally, then a serum glucose will be obtained 2 hours later. Serum glucose is measured in mg/dL.

SECONDARY OUTCOMES:
Change in serum insulin levels during a glucose tolerance test | Baseline, twelve weeks
  Serum insulin levels in multi-international units per litre (mIU/L) will be measured at baseline and after 2 hours during a 2-hour glucose tolerance test
Serum Testosterone | Baseline, twelve weeks
  Serum testosterone in ng/dL Changes in serum testosterone as measured in ng/dL
Sex hormone binding globulin | Baseline, twelve weeks
  Changes in sex hormone binding globulin in nmol/L
Stool sample | Baseline, twelve weeks
  Gut microbiota
Inflammatory marker cluster of differentiation 4 (CD4) | Baseline, twelve weeks
  CD4
Inflammatory marker cluster of differentiation 8 (CD8) | Baseline, twelve weeks
  CD8
Inflammatory marker Foxp3 | Baseline, twelve weeks
  Foxp3
Inflammatory marker cluster of differentiation 11b (CD11b) | Baseline, twelve weeks
  CD11b
Inflammatory marker cluster of differentiation 33 (CD33) | Baseline, twelve weeks
  CD33
Inflammatory marker F4/80 | Baseline, twelve weeks
  F4/80
Inflammatory marker interleukin 10 (IL-10) | Baseline, twelve weeks
  IL-10
Inflammatory marker interleukin 1b (IL-1b) | Baseline, twelve weeks
  IL-1b
Inflammatory marker tumor necrosis factor alpha (TNF-a) | Baseline, twelve weeks
  TNF-a
Inflammatory marker interleukin 6 (IL-6) | Baseline, twelve weeks
  IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Henry Bohler, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States